CLINICAL TRIAL: NCT00657267
Title: Phase 2 Study of Dose-Intense Temozolomide in Recurrent Glioblastoma
Brief Title: Dose-Intense Temozolomide in Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Y. Wen, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); University of Pennsylvania (Other); Wake Forest University Health Sciences (Other); Tufts Medical Center (Other); Dartmouth-Hitchcock Medical Center (Other); Schering-Plough (Industry)
Responsible Party: Sponsor-Investigator, Patrick Y. Wen, MD, Director, Center for Neuro-Oncology, Dana-Farber Cancer Institute, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-013; P05516 (Other: Schering Plough)
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: recurrent glioblastoma; temodar; temozolomide
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-Arm Study (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Taken orally daily for the first three weeks of a four-week cycle.
  Other Names: Temodar

SUMMARY:
Temozolomide (Temodar) is an FDA approved medication for the treatment of newly diagnosed glioblastomas. In this study, we will be using temozolomide to treat recurrent glioblastomas. We will be using a different dose and schedule than the FDA approved dose and schedule. The purpose of this study is to determine if patients that have failed standard temozolomide treatment will respond to temozolomide when given at a different dose and schedule (21 days every 28 days).

DETAILED DESCRIPTION:
* Participants will be given a medication-dosing calendar for each treatment cycle. Each treatment cycle lasts 4 weeks (28 days) during which time they will be taking temozolomide orally once a day for the first three weeks.
* At the end of each cycle (day 28, +/- 2 days), the following procedures will be performed: Complete physical examination including a neurological exam; vital signs; a review of current medications and symptoms; blood samples; a pregnancy test for women of child-bearing potential; self-administered quality of life questionnaire; brain MRI or CT scan.
* Participants may continue taking temozolomide until their tumor grows or if they experience unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must provide independent consent or must demonstrate willingness to participate in the study and to adhere to dose and visit schedules.
* 18 years of age or older (of either sex, and of any race)
* Histologic diagnosis of GBM or gliosarcoma with an unequivocal progression by MRI or CT scan
* Must have received standard combined modality therapy as first-line treatment consisting of RT plus concomitant temozolomide followed by adjuvant temozolomide (at least 2 cycles of adjuvant temozolomide)
* Gadolinium MRI or contrast CT scan must be obtained within 14 days prior to registration, and must be on a steroid dose that has been stable for at least 5 days.
* Karnofsky Performance status of 60 or greater
* Life expectancy of at least 8 weeks
* Recovered from the toxic effects of prior therapy, and 21 days must have elapsed since prior treatment with temozolomide

  o If a patient has residual toxicity from any previous treatment, toxicity must be ≤ Grade 1
* Laboratory tests within parameters outlined in the protocol
* Female subjects of childbearing potential & male subjects with female partner of childbearing potential must agree to use a medically accepted method of contraception or be surgically sterilized prior to Screening, while receiving protocol-specified medication, and for 30 days after stopping the study medication
* Negative pregnancy test within 48 hours prior to dosing with the study drug (for female subjects of childbearing potential)
* Free of any clinically relevant disease that would, in the Principal Investigator's opinion, interfere with the conduct of the study or study evaluations
* Must be able to adhere to the dosing and visit schedules, and agree to record medication times, concomitant medications, and adverse events (AEs) accurately and consistently in a daily diary
* Unstained slides (at least 15 of 10 micron thickness, or 20 when < 10 micron thickness)or 1 tissue block must be available from the original diagnostic biopsy/surgery or from the biopsy/surgery recurrence
* Participants who have undergone recent resection of recurrent or progressive tumor will be eligible provided at least 2 weeks has elapsed since surgery, and subjects have recovered from surgical-related trauma
* Residual disease following resection of recurrent GBM or gliosarcoma is not mandated for eligibility into the study.

Exclusion Criteria:

* Participant has received a dosing schedule of temozolomide other than 75 mg/m2/day for 42 days during RT followed by adjuvant temozolomide at a dose of 150-200 mg/m2/day for 5 days of a 28-day schedule (standard dose adjustments for toxicity are allowed)
* Any other anti-tumor agent other than standard surgical resection, RT and temozolomide prior to enrollment or during the study period
* Received treatment with BCNU (Gliadel) wafers or GliaSite
* Progressed prior to receiving at least 2 cycles of adjuvant temozolomide
* Pregnant or intending to become pregnant during the study
* In a situation or condition that, in the opinion of the Investigator, may interfere with optimal participation in the study
* Participating in any other clinical study in which an investigational drug is prescribed
* Allergic to or has sensitivity to the study drug or its excipients
* History of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless he/she is in complete remission and has not received treatment for that particular disease for the past 3 or more years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-05; Primary Completion 2011-11 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Wake Forest Univsersity, Winston-Salem, North Carolina
  - University Of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study activated at DFCI in May 2008 and was eventually activated at MGH, UPENN, Wake Forest University Baptist Medical Center, Dartmouth-Hitchcock Medical Center, and Tufts NEMC.
Groups:
- 12 Cycles of Dose-Dense Temozolomide (Single Arm Study): Temozolomide dose = 100 mg/m2/day for 21 days of every 28-day cycle (75 mg/m2/day for 21 days of every 28-day cycle if pt experienced myelosuppression on prior regimen: gr 1 ANC &/or gr 2 platelets)
Period: Overall Study
Arm/Group | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study)
Started | 58
Completed | 4
Not Completed | 54
Not completed — Progressive disease | 45
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Population: Of the 58 participants who registered and started study treatment, 3 were ineligible for analysis and 1 withdrew before response assessment.
Arm/Group | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study)
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 57 [25 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 51
  More than one race | 2
  Unknown or Not Reported | 3
Karnofsky performance status (KPS) at registration [Median (Full Range); unit: %] — KPS scores:
  100% normal 90% normal activity; minor signs or symptoms 80% normal activity w/ effort; some signs or symptoms 70% cares for self; unable to do normal activity or active work 60% requires occasional assistance, but cares for most personal needs 50% requires considerable assistance and frequent medical care 40% disabled; requires special care and assistance 30% severely disabled; hospital admission is indicated but death not imminent 20% very sick; hospitalization necessary; active supportive treatment necessary 10% moribund; fatal processes progressing rapidly 0% dead
  % | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival
Description: Progression is defined using Modified Macdonald Criteria , using a >/= 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR clear clinical worsening or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months
Population: Patients evaluable for imaging analysis, as protocol-defined.
Measure: Number; unit: percentage of evaluable participants
Arm/Group | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study)
Number analyzed (Participants) | 55
percentage of evaluable participants | 11

2. Secondary Outcome: Overall Survival
Time Frame: From patient registration until end of study, assessed up to 54 months
Population: Entire study population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study)
Number analyzed (Participants) | 58
months | 11.7 [8.1 to 16.2]

3. Secondary Outcome: Radiographic Response
Description: Responders on study are those with a best response of either CR or PR. Per Modified Macdonald Criteria for lesions assessed by MRI/CT: Complete Response (CR) = Complete disappearance of all measurable and evaluable disease, no new lesions, no evidence of non-evaluable disease, with no steroids. Partial Response (PR) >/= 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions, no progression of evaluable disease, no new lesions, with steroid dose @ time of response </= max dose w/in the first 8 weeks of therapy.
Time Frame: From patient registration until end of study, assessed up to 54 months
Population: Of the 58 patients registered, 3 of were ineligible for analysis based on path review, which is why only 55 patients were evaluated for this outcome.
Measure: Number; unit: percentage of participants evaluated
Groups:
- Partial Response: Partial Responders on study; Temozolomide dose = 100 mg/m2/day for 21 days of every 28-day cycle (75 mg/m2/day for 21 days of every 28-day cycle if pt experienced myelosuppression on prior regimen: gr 1 ANC &/or gr 2 platelets)
- Complete Response: Complete responders on study; Temozolomide dose = 100 mg/m2/day for 21 days of every 28-day cycle (75 mg/m2/day for 21 days of every 28-day cycle if pt experienced myelosuppression on prior regimen: gr 1 ANC &/or gr 2 platelets)
Arm/Group | Partial Response | Complete Response
Number analyzed (Participants) | 55 | 55
percentage of participants evaluated | 13 | 0

4. Secondary Outcome: Time to Progression.
Description: as for outcome 1
Time Frame: From patient registration until end of study, assessed up to 54 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study)
Number analyzed (Participants) | 55
days | 56 [56 to 84]

ADVERSE EVENTS:
Time Frame: SAEs are reported from the signing of the consent form until the 30-Days-After-Last Dose-of Study Drug Visit. (Any SAEs occurring within the 30 days after last dose of study drug need to be followed until resolved.)
Description: AEs collected via regular Investigator assessment and regular laboratory testing.
Groups:
- 12 Cycles of Dose-Dense Temozolomide (Single Arm Study): All 58 participants who started treatment: Temozolomide dose = 100 mg/m2/day for 21 days of every 28-day cycle (75 mg/m2/day for 21 days of every 28-day cycle if pt experienced myelosuppression on prior regimen: gr 1 ANC &/or gr 2 platelets
Arm/Group | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study)
Serious Adverse Events (participants affected / at risk) | 19/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study) (N=58)
Disease Progression NOS (General disorders) | 2 (2) — Death due to progressive disease within 30 days of last dose of study drug
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Seizure (Nervous system disorders) | 6 (6)
Neurology - Other (Nervous system disorders) | 2 (2) — Hospital admission for progressive disease (craniotomy, etc.)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 (1) — Hospital admission for methemoglobinemia (Dapsone-induced)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 7 (18)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1)
Speech impairment (Nervous system disorders) | 2 (2)
Muscle weakness - left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) — with a fall
Supraventricular and nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 1 (1)
Pain - headache (Nervous system disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (4)
Vomiting (Gastrointestinal disorders) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 1 (4)
Distension/bloating, (Gastrointestinal disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Potassium, serum-low (Hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Pain - Chest NOS (General disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2 (3) — Hospitilization for Mechanical Fall
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12 Cycles of Dose-Dense Temozolomide (Single Arm Study) (N=58)
Hemoglobin (Blood and lymphatic system disorders) | 25
Leukocytes (Blood and lymphatic system disorders) | 34
Lymphopenia (Blood and lymphatic system disorders) | 49
Neutrophils (Blood and lymphatic system disorders) | 17
Platelets (Blood and lymphatic system disorders) | 30
INR (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 41
Insomnia (General disorders) | 10
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Cushingnoid appearance (Endocrine disorders) | 5
Anorexia (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 19
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 4
Incontinence- anal (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 7
Edema limb (Blood and lymphatic system disorders) | 13
Alkaline phosphatase (Metabolism and nutrition disorders) | 7
ALT- SGPT (Metabolism and nutrition disorders) | 14
AST- SGOT (Metabolism and nutrition disorders) | 13
Bicarbonate (Metabolism and nutrition disorders) | 10
Bilirubin (Metabolism and nutrition disorders) | 8
Creatinine (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 39
Hyperkalemia (Metabolism and nutrition disorders) | 12
Hypernatremia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Proteinuria (Metabolism and nutrition disorders) | 3
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 14
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 7
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 6
Nonneuropathic right-side muscle weak (Musculoskeletal and connective tissue disorders) | 3
Anxiety (Nervous system disorders) | 6
Ataxia (Nervous system disorders) | 4
Cognitive disturbance (Nervous system disorders) | 5
Confusion (Nervous system disorders) | 15
Depressed level of consciousness (Nervous system disorders) | 3
Depression (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 9
Memory impairment (Nervous system disorders) | 22
Neuropathy CN II vision (Nervous system disorders) | 5
Neuropathy CN VII face-motor / taste (Nervous system disorders) | 6
Neuropathy CN VIII hearing & balance (Nervous system disorders) | 6
Neuropathy-motor (Nervous system disorders) | 22
Neuropathy-sensory (Nervous system disorders) | 14
Seizure (Nervous system disorders) | 11
Speech impairment (Nervous system disorders) | 17
Tremor (Nervous system disorders) | 4
Cataract (Eye disorders) | 3
Vision-blurred (Eye disorders) | 8
Abdomen- pain (Gastrointestinal disorders) | 3
Back- pain (Musculoskeletal and connective tissue disorders) | 5
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 4
Head/headache (Nervous system disorders) | 24
Joint- pain (Musculoskeletal and connective tissue disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3
Incontinence urinary (Renal and urinary disorders) | 10
Urinary frequency/urgency (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days